CLINICAL TRIAL: NCT02822170
Title: A Pilot Study of Combined Cycle Ergometry and Amino Acids in the ICU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont (Other)
Responsible Party: Principal Investigator, Renee Stapleton, Associate Professor of Medicine, University of Vermont
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHRMS16-540
Record Dates: First submitted 2016-06-25; First posted 2016-07-04 (Estimated); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Acute Respiratory Failure
MeSH Terms: interventions — Amino Acids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IV amino acids and in-bed cycle ergometry (Experimental): Beginning within 96 hours of ICU admission, participants will receive the following combined intervention:
  1. IV amino acids (15% solution) delivered by continuous infusion, such that the total enteral and IV protein will be between 2.0-2.5 g/kg/day.
  2. In-bed cycle ergometry exercise delivered in 45-minute sessions 5 days per week according to a detailed specific protocol that includes a safety check and gradual increases in resistance if the participant is actively cycling.
  Interventions: Other: IV amino acids and in-bed cycle ergometry

INTERVENTIONS:
Other: IV amino acids and in-bed cycle ergometry — IV amino acids and in-bed cycle ergometry

SUMMARY:
The purpose of this small pilot study is to refine a combined intervention of IV amino acids and cycle ergometry in critically ill patients, and to gather preliminary data, before proceeding with a larger multi-center RCT. A total of 10 patients will receive the combined intervention.

ELIGIBILITY:
Inclusion Criteria:

1. >=18 years old
2. Requiring mechanical ventilation or high flow nasal cannula (HFNC) with actual or expected total duration of mechanical ventilation or HFNC >48 hours
3. Expected ICU stay >4 days after enrollment (to permit adequate exposure to the proposed intervention)

Exclusion Criteria:

1. >120 continuous hours of mechanical ventilation or HFNC before enrollment
2. Expected death or withdrawal of life-sustaining treatments within 7 days from enrollment
3. No expectation for any nutritional intake within the subsequent 72 hours
4. Severe chronic liver disease (MELD score >20) or acute fulminant hepatitis.
5. Documented allergy to the amino acid intervention
6. Not ambulating independently prior to ICU admission (use of gait aid permitted)
7. Pre-existing primary systemic neuromuscular disease (e.g. Guillain Barre)
8. Neuromuscular blocker infusion (eligible once infusion discontinued if other inclusion criteria met)
9. Pre-existing intracranial or spinal process affecting motor function
10. Pre-existing cognitive impairment or language barrier that prohibits outcomes assessment
11. Lower extremity impairments that prevent cycling (e.g. amputation, knee/hip injury)
12. Weight >150kg
13. Pregnant
14. Incarcerated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
6-minute walk distance (6MWD) | 6MWD will be measured near the time that the particioant is being discharged from the hospital, up to 26 weeks after randomization.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Vermont College of Medicine, Burlington, Vermont, United States